CLINICAL TRIAL: NCT07005128
Title: A Phase 3, Open Label, Multicenter, Randomized Study of First Line Tarlatamab in Combination With Durvalumab, Carboplatin and Etoposide Versus Durvalumab, Carboplatin and Etoposide in Untreated Extensive Stage Small-Cell Lung Cancer (DeLLphi-312)
Brief Title: A Study Comparing Tarlatamab, Durvalumab, Carboplatin, and Etoposide Versus Durvalumab, Carboplatin, and Etoposide in First-line Extensive Stage Small-Cell Lung Cancer (ES-SCLC)
Acronym: DeLLphi-312
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20240178
Record Dates: First submitted 2025-05-27; First posted 2025-06-05 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Small-cell Lung Cancer; Extensive Stage Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — AMG 757; durvalumab; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tarlatamab + Durvalumab + Carboplatin + Etoposide (Experimental): Participants will receive tarlatamab in combination with durvalumab, carboplatin and etoposide for 4 cycles followed by tarlatamab and durvalumab.
  Interventions: Drug: Tarlatamab; Drug: Durvalumab; Drug: Carboplatin; Drug: Etoposide
- Durvalumab + Carboplatin + Etoposide (Active Comparator): Participants will receive durvalumab, carboplatin and etoposide for 4 cycles followed by durvalumab.
  Interventions: Drug: Durvalumab; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Tarlatamab — Tarlatamab will be administered as an intravenous (IV) infusion.
  Other Names: AMG 757; Imdelltra
  Arms: Tarlatamab + Durvalumab + Carboplatin + Etoposide
Drug: Durvalumab — Durvalumab will be administered as an IV infusion.
Drug: Carboplatin — Carboplatin will be administered as an IV infusion.
Drug: Etoposide — Etoposide will be administered as an IV infusion.

SUMMARY:
The main objective of the study is to compare the efficacy of tarlatamab in combination with durvalumab, carboplatin and etoposide to the combination of durvalumab, carboplatin and etoposide on prolonging overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* Participant has provided informed consent before initiation of any study-specific activities/procedures.
* Age ≥ 18 years or ≥ legal age within the country if it is older than 18 years.
* Histologically or cytologically documented ES-SCLC (American Joint Committee on Cancer, 2017, Stage IV SCLC [T any, N any, M1 a/b/c]), or T3 to T4 due to multiple lung nodules that are too extensive or have tumor/nodal volume that is too large to be encompassed in a tolerable radiation plan.
* Measurable disease as defined per RECIST 1.1.
* Suitable to receive carboplatin, etoposide and durvalumab regimen as first-line treatment per investigator clinical assessment.
* Minimum life expectancy ≥ 12 weeks.

Exclusion Criteria:

* Participants can have no history of other malignancy in the last 2 years.
* Any symptomatic central nervous system (CNS) metastases, or leptomeningeal disease.
* They will have no history of severe or life-threatening events to immune-mediated therapy.
* History of arterial thrombosis (eg, stroke or transient ischemic attack) within 6 months prior to first dose of study treatment.
* They will have no active autoimmune or inflammatory disorders.
* Presence of active human immunodeficiency virus (HIV) or active Hepatitis (B/C) infection.
* Evidence or interstitial lung disease (ILD) or active, non-infectious pneumonitis.
* History of solid organ transplant.
* They will not have had a myocardial infarction and/or symptomatic congestive heart failure (New York Heart Association > class II) within 6 months prior to first dose of study treatment.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2029-01-04 (Estimated); Study Completion 2029-07-15 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to approximately 3.5 years
Progression free survival (PFS) (Blinded Independent Central Review [BICR] Assessed) | Up to approximately 3.5 years

SECONDARY OUTCOMES:
PFS (Investigator Assessed) | Up to approximately 4 years
Objective Response (OR) | Up to approximately 4 years
Disease Control | Up to approximately 4 years
Duration of Response (DOR) | Up to approximately 4 years
PFS Rate | 6 months, 1 year, and 2 years
OS Rate | 6 months, 1 year, 2 years and 3 years
Time to Progression | Up to approximately 4 years
Number of Participants Who Experience Treatment-emergent Adverse Events (TEAEs) | Up to approximately 4 years
Number of Participants Who Experience Treatment-related Adverse Events | Up to approximately 4 years
Number of Participants Who Experience Events of Interest | Up to approximately 4 years
Serum Concentrations of Tarlatamab | Up to approximately 1 year
Number of Participant Who Develop Anti-Tarlatamab Antibodies | Up to 13 months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (119):
- United States (12):
  - Saint Bernards Medical Center, Jonesboro, Arkansas
  - Presbyterian Intercommunity Hospital Health Whitter Hospital, Whittier, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - University of Illinois Chicago, Chicago, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Cancer Center of Kansas, Heritage Plaza Medical Building, Wichita, Kansas
  - Allina Health System dba Allina Health Cancer Institute, Minneapolis, Minnesota
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Kaiser Permanente Medical Center, Portland, Oregon
  - Baptist Cancer Center, Memphis, Tennessee
  - Swedish Cancer Institute Medical Oncology, Seattle, Washington
  - West Virginia University Health Sciences Center, Morgantown, West Virginia
- Argentina (3):
  - Cemic, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital Universitario Austral, Pilar, Buenos Aires
  - Sanatorio Parque SA, Rosario, Santa Fe Province
- Australia (2):
  - Chris OBrien Lifehouse, Camperdown, New South Wales
  - Monash Medical Centre, Clayton, Victoria
- Austria (2):
  - Medizinische Universitaet Graz, Graz
  - Universitaetsklinikum Krems, Krems
- Belgium (4):
  - Jessa Ziekenhuis - Campus Virga Jesse, Hasselt
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven
  - AZ Delta Campus Rumbeke, Roeselare
  - Centre Hospitalier Universitaire-Universite Catholique de Louvain Namur-Site Godinne, Yvoir
- Brazil (4):
  - Cenantron Centro Avançado de Tratamento Oncologico Ltda, Belo Horizonte, Minas Gerais
  - Liga Norte-Riograndense Contra O Cancer, Natal, Rio Grande do Norte
  - Hospital Sao Lucas da Pontificia Universidade Catolica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Fund Faculdade Regional Med Sao Jose Rio Preto, São José do Rio Preto, São Paulo
- China (17):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - The Second Attached Hospital Of Fujian Medical University, Quanzhou, Fujian
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Jiamusi Cancer Hospital, Jiamusi, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Jiangxi Cancer hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shandong Cancer Hospital, Jinan, Shandong
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - Tianjin Peoples Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital Of Ningbo University, Ningbo, Zhejiang
  - Beijing Cancer Hospital, Beijing
  - Fujian Cancer Hospital, Fuzhou
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Regionshospitalet Godstrup, Herning
- France (7):
  - Centre Hospitalier Intercommunal de Creteil, Créteil
  - Centre Leon Berard, Lyon
  - Centre Hospitalier Universitaire Nord, Marseille
  - Institut Curie, Paris
  - Centre Hospitalier Universitaire de Nantes - Hopital Nord Laennec, Saint-Herblain
  - Hopital d instruction des armees sainte anne, Toulon
  - Centre Hospitalier Universitaire de Toulouse - Hopital Larrey, Toulouse
- Germany (9):
  - Klinikum Chemnitz GmbH, Chemnitz
  - Krankenhaus Koeln-Merheim - Kliniken der Stadt Koeln gGmbH, Cologne
  - Universitaetsklinikum Dresden, Dresden
  - Krankenhaus Nordwest, Frankfurt am Main
  - Asklepios Fachkliniken Muenchen Gauting, Gauting
  - LungenClinic Grosshansdorf GmbH, Großhansdorf
  - Universitaetsklinikum Schleswig-Holstein - Kiel, Kiel
  - Universitaetsklinikum Schleswig-Holstein - Luebeck, Lübeck
  - Universitaetsklinikum Wuerzburg, Würzburg
- Greece (4):
  - Henry Dunant Hospital Center, Athens
  - Alexandra Hospital, Athens
  - European Interbalkan Medical Center, Thessaloniki
  - Iatriko Diavalkaniko Thessalonikis, Thessaloniki
- Hong Kong (2):
  - Queen Mary Hospital, The University of Hong Kong, Hong Kong
  - Prince of Wales Hospital, Chinese University of Hong Kong, Shatin, New Territories
- Hungary (2):
  - Matrai Gyogyintezet, Gyöngyös
  - Reformatus Pulmonologiai Centrum, Törökbálint
- Italy (6):
  - IRCCS Istituto Tumori Giovanni Paolo II, Bari
  - Humanitas Gavazzeni, Bergamo
  - Istituto Romagnolo per lo Studio dei Tumori Dino Amadori, Meldola (FC)
  - IRCCS Istituto Oncologico Europeo, Milan
  - Azienda Ospedaliera San Giovanni Addolorata, Roma
  - Centro Ricerche Cliniche Di Verona Societa responsabilita limitata, Verona
- Japan (13):
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi-shi, Hyōgo
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Okayama University Hospital, Okayama, Okayama-ken
  - Kansai Medical University Hospital, Hirakata-shi, Osaka
  - Osaka International Cancer Institute, Osaka, Osaka
  - Kindai University Hospital, Sakai-shi, Osaka
  - Saitama Medical University International Medical Center, Hidaka-shi, Saitama
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - Wakayama Medical University Hospital, Wakayama, Wakayama
- Netherlands (3):
  - Universitair Medisch Centrum Groningen, Groningen
  - Maastricht Universitair Medisch Centrum, Maastricht
  - Erasmus Medisch Centrum, Rotterdam
- Poland (2):
  - Centrum Pulmonologii i Torakochirurgii w Bystrej, Bystra
  - Instytut Gruzlicy i Chorob Pluc, Warsaw
- Portugal (3):
  - Hospital Cuf Tejo, Lisbon
  - Hospital da Luz, SA, Lisbon
  - Unidade Local de Saude de Matosinhos, EPE - Hospital Pedro Hispano, Matosinhos Municipality
- Institutul Oncologic Prof Dr Ion Chiricuta Cluj-Napoca, Cluj-Napoca, Romania
- South Korea (3):
  - Chungbuk National University Hospital, Cheongju Chungbuk
  - National Cancer Center, Goyang-si Gyeonggi-do
  - Severance Hospital Yonsei University Health System, Seoul
- Spain (7):
  - Hospital Regional Universitario de Malaga, Málaga, Andalusia
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital Universitari i Politecnic La Fe, Valencia, Valencia
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Switzerland (3):
  - Universitaetsspital Basel, Basel
  - Kantonsspital Graubuenden, Chur
  - Hopitaux universitaires de Geneve, Geneva
- Taiwan (2):
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
- Turkey (Türkiye) (6):
  - Memorial Ankara Hastanesi, Ankara
  - Ankara Bilkent Sehir Hastanesi, Ankara
  - Bagcilar Medipol Mega Universite Hastanesi, Istanbul
  - Goztepe Prof Dr Suleyman Yalcin Sehir Hastanesi, Istanbul
  - Ege Universitesi Tip Fakultesi Hastanesi, Izmir
  - Sakarya Egitim ve Arastirma Hastanesi, Sakarya

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com